CLINICAL TRIAL: NCT02562352
Title: Team Approach to Polypharmacy Evaluation and Reduction: Feasibility Study
Brief Title: Team Approach to Polypharmacy Evaluation and Reduction
Acronym: TAPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Health Canada (Other Government); The Labarge Optimal Aging Initiative (Other); David Braley and Nancy Gordon Chair in Family Medicine (Other); RxISK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TAPER-001-19-Aug-15
Record Dates: First submitted 2015-08-21; First posted 2015-09-29 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Comorbidity; Medication Therapy Management
Keywords: polypharmacy; multimorbidity; randomized controlled trial; drug discontinuation; patient preference; eHealth
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAPER program (Experimental): The intervention arm is comprised of:
  1. Identification of medications that are appropriate for discontinuation/dose reduction.
  2. Linked pharmacist/family physician consultations with patient to discuss medication discontinuation/dose reduction.
  Interventions: Other: TAPER program
- Control (No Intervention): Standard of Care as wait list control

INTERVENTIONS:
Other: TAPER program — Patients will be randomized to receive the TAPER program at study start or delayed intervention at 6 months.
  Other Names: Medication Discontinuation/Dose Reduction
  Arms: TAPER program

SUMMARY:
In an aging population, most seniors suffer from multiple chronic conditions. When the number of medications taken is ≥5 (polypharmacy), the burden of taking so many together can do more harm than good. This study will test a program focused on medication reduction involving patient, pharmacist and physician using current technology aimed at reducing the harms of polypharmacy. Reducing the risk of adverse effects from drugs or the interactions between them involves prioritizing the most important ones according to the patient's preference and stopping those which may no longer be necessary. Reducing the dose also reduces the risk of drug side effects. Patients, aged over 69 years taking ≥5 medications, will randomly receive the program immediately or at 6 months. The program involves information gathering from the patient, medication review with the pharmacist and then a consultation with the family doctor focused on discontinuing/reducing the dose of medications where possible using a 'pause and monitor' framework to assess the need for restart. An electronic program that detects drug adverse effects and flags potentially inappropriate medications will be integrated into a clinical pathway incorporating monitoring and follow up systems. This study will examine effects on patient and health relevant outcome measures as well as patients' and clinicians' experiences of the program. The results will be used to determine whether this system can be implemented as part of routine preventative care in older adults.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to receive the intervention at study start or delayed appointment 6 months later. The intervention includes initial baseline data collection from the patient including data on demographics, medications, and illness characteristics. The patient will then attend an appointment with a pharmacist to review medications appropriate for discontinuation/dose reduction, after which the patient will meet with his/her family physician to discuss patient preferences for discontinuation/dose reduction. Follow up appointments will take place at one week, 3 months and 6 months (study end). Questionnaires and a semi-structured interview will take place at the 6 month appointment. After six months, the control group will be offered the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years of age or older
* Participating family doctor as most responsible provider
* Patient of McMaster Family Health Team
* Currently taking 5 or more medications
* Have not had a recent comprehensive medication review
* Patient consents

Exclusion Criteria:

* English language or cognitive skills inadequate to understand and respond to rating scales
* Terminal illness or other circumstance precluding 13 month study period

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Successful discontinuation (Difference in mean number of medications) | 6 months
  Difference in mean number of medications per patient.

SECONDARY OUTCOMES:
Quality of Life (EQ-5D) | 6 months
  EQ-5D
Nutritional Status (Mini Nutritional Assessment Short-Form) | 6 months
  Mini Nutritional Assessment Short-Form;
Patient experience of deprescribing (Thematic analysis of semi structured interviews) | 6 months
  Thematic analysis of semi structured interviews
Physical Functional Capacity (Manty structured validated interview) | 6 months
  Manty structured validated interview
Falls (self report number of falls) | 6 months
  self report number of falls
Adverse Events (patient self report or clinician report) | 6 months
  patient self report or clinician report
Health Resource Utilization (Number of hospital admissions and emergency dept visits) | 6 months
  Number of hospital admissions and emergency dept visits
Cognition (The Mini Mental Status Examination) | 6 months
  The Mini Mental Status Examination
Fatigue (Avlund Mob-T Scale) | 6 months
  Avlund Mob-T Scale
Patient Enablement (Patient Enablement Index) | 6 months
  Patient Enablement Index
Self-Efficacy (Stanford Self-Efficacy Scale) | 6 months
  Stanford Self-Efficacy Scale
Patient self report of change in quality of life/morbidity (Global Impression Scale) | 6 months
  Global Impression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Dee Mangin, MBChB, DPH, FRNZC, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Mangin D, Lamarche L, Agarwal G, Ali A, Cassels A, Colwill K, Dolovich L, Brown ND, Farrell B, Freeman K, Frizzle K, Garrison SR, Gillett J, Holbrook A, Jurcic-Vrataric J, McCormack J, Parascandalo J, Richardson J, Risdon C, Sherifali D, Siu H, Borhan S, Templeton JA, Thabane L, Trimble J. Team approach to polypharmacy evaluation and reduction: feasibility randomized trial of a structured clinical pathway to reduce polypharmacy. Pilot Feasibility Stud. 2023 May 18;9(1):84. doi: 10.1186/s40814-023-01315-0. PMID 37202822